CLINICAL TRIAL: NCT04845217
Title: Efficacy of Peppermint Oil in a Randomized, Single-Blind, Placebo Controlled Trial in Women With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Peppermint Oil for the Treatment of Interstitial Cystitis / Bladder Pain Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Integrative Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Sean Francis, MD, Professor, MD, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21.0286
Record Dates: First submitted 2021-03-29; First posted 2021-04-14 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Interstitial Cystitis
Keywords: interstitial cystitis; bladder pain syndrome; peppermint
MeSH Terms: conditions — Cystitis, Interstitial | interventions — peppermint oil; Coconut Oil

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to the intervention or placebo arm. Allocation concealment will be in place to ensure the individual enrolling the subject into the study has no a priori knowledge of group assignment. Block randomization will occur with randomly mixed block sizes of 4, 6, and 8 using the randomization list generator at www.sealedenvelope.com. Randomization information will be kept confidential and only available to study personnel.
Who Masked: Participant
Masking Description: The peppermint-oil and placebo treatments will be kept in a locked and secured area of the office, in a room not used for patient care. The bottles will be de-identified, with labels detailing the specific instructions for how to take the soft gels and the number in each bottle. Each group will be instructed to take one soft gel three times daily.
  The peppermint oil and placebo medications will be distributed by the research team. The manufacturer label will be covered up/removed and a study label stating the use of a study medication will be used to maintain patient blinding.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Peppermint Oil (Experimental): Participants in the intervention (peppermint oil) arm will receive soft gels of enteric-coated peppermint oil (0.2mL=200mg). The enteric coated peppermint oil soft gel utilized in this study is Peptogest Peppermint Oil from Schwabe North America (Nature's Way Brand).
  Interventions: Drug: Peppermint oil
- Coconut Oil (Placebo Comparator): Participants in the placebo (coconut oil) arm will receive soft gels of enteric coated coconut oil. The enteric coated coconut oil soft gel utilized in this study is Coconut Oil from Schwabe North America (Nature's Way Brand).
  Interventions: Drug: Coconut Oil

INTERVENTIONS:
Drug: Peppermint oil — Enteric coated peppermint oil taken by mouth three times daily for 8 weeks.
  Other Names: Peptogest Peppermint Oil
  Arms: Peppermint Oil
Drug: Coconut Oil — Enteric coated coconut oil taken by mouth three times daily for 8 weeks
  Other Names: Coconut Oil Pure Extra Virgin
  Arms: Coconut Oil

SUMMARY:
The purpose of this study is to assess the use of peppermint oil as a treatment for Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS).

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants will complete validated IC/BPS symptom questionnaires for baseline screening. Once participants meet eligibility requirements and give written informed consent they will be randomized in a 1:1 ratio to peppermint oil (200mg TID) or placebo (also TID). Participants will complete validated IC/BPS questionnaires and follow up surveys over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-65 years old
* Diagnosed with IC/BPS for at least one month prior to study enrollment

Exclusion Criteria:

* Culture proven urinary tract infection within 1 month of randomization
* Gross hematuria
* Currently pregnant or breastfeeding
* Unable to speak and read English
* History of allergic reaction to peppermint, coconut or enteric coating
* History of malabsorption syndrome
* History of gastroparesis
* History of gastric bypass surgery
* History of gastrointestinal, genitourinary or pelvic cancer in the last 5 years
* History of insulin dependent diabetes
* History of active urinary stone disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
O'Leary/Sant questionnaire scores | 8 weeks
  Participant responses to the O'Leary/Sant questionnaire assessing IC/BPS symptoms will be compared at baseline and after starting treatment with peppermint oil.
Pelvic Pain and Urgency/Frequency questionnaire scores | 8 weeks
  Participant responses to the Pelvic Pain and Urgency/Frequency questionnaire assessing IC/BPS symptoms will be compared at baseline and after starting treatment with peppermint oil.

SECONDARY OUTCOMES:
Urine pH | 8 weeks
  Changes in urine pH on urine dipstick from clinically indicated lab collections at the time of office visits during the study period
Incidence of urinary tract infections (UTIs) | 8 weeks
  Culture proven UTIs during the study period (>100,000 CFU of a single pathogen)
Additional IC/BPS Treatments received | 8 weeks
  Number and type of additional IC/BPS each participant undergoes

CONTACTS AND LOCATIONS:
Overall Officials: Sean Francis, MD, Principal Investigator — Department Chair
Locations (1):
- Springs Medical Center, Louisville, Kentucky, United States